CLINICAL TRIAL: NCT00168454
Title: A Research Study for Patients With Overactive Bladder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191622-077
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2010-02-11 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-10

CONDITIONS: Overactive Bladder; Urinary Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo (Placebo Comparator): Placebo (normal saline) injected into detrusor on Day 1
  Interventions: Drug: Placebo
- BOTOX 50 U (Experimental): botulinum toxin Type A 50 U injected into detrusor on Day 1
  Interventions: Biological: botulinum toxin Type A
- BOTOX 100 U (Experimental): botulinum toxin Type A 100 U injected into detrusor on Day 1
  Interventions: Biological: botulinum toxin Type A
- BOTOX 150 U (Experimental): botulinum toxin Type A 150 U injected into detrusor on Day 1
  Interventions: Biological: botulinum toxin Type A
- BOTOX 200 U (Experimental): botulinum toxin Type A 200 U injected into detrusor on Day 1
  Interventions: Biological: botulinum toxin Type A
- BOTOX 300 U (Experimental): botulinum toxin Type A 300 U injected into detrusor on Day 1
  Interventions: Biological: botulinum toxin Type A

INTERVENTIONS:
Biological: botulinum toxin Type A — botulinum toxin Type A injected into detrusor on Day 1
  Other Names: BOTOX®
  Arms: BOTOX 100 U; BOTOX 150 U; BOTOX 200 U; BOTOX 300 U; BOTOX 50 U
Drug: Placebo — Placebo (normal saline) injected into detrusor on Day 1
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate whether injections of botulinum toxin Type A into the bladder are safe and effective in treating overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18-85 years old
* Must have been diagnosed by his/her doctor with overactive bladder at least 6 months ago
* Must weigh at least 50 kg (110 lbs)
* Must be willing and able to record information regarding bladder function into a diary (provided)
* Must be willing and able to complete the entire course of the study

Exclusion Criteria:

* Cannot currently be catheterizing as a way to control incontinence
* Must not have used botulinum toxin type A or any other botulinum toxin previously for any condition

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2005-07; Primary Completion 2008-01 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (6):
- Pittsburgh, Pennsylvania, United States
- Ghent, Belgium
- Victoria, British Columbia, Canada
- Berlin, Germany
- Warsaw, Poland
- Sheffield, United Kingdom

REFERENCES:
- [Derived] Fowler CJ, Auerbach S, Ginsberg D, Hale D, Radziszewski P, Rechberger T, Patel VD, Zhou J, Thompson C, Kowalski JW. OnabotulinumtoxinA improves health-related quality of life in patients with urinary incontinence due to idiopathic overactive bladder: a 36-week, double-blind, placebo-controlled, randomized, dose-ranging trial. Eur Urol. 2012 Jul;62(1):148-57. doi: 10.1016/j.eururo.2012.03.005. Epub 2012 Mar 14. PMID 22464310

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo (normal saline)injection on Day 1 into detrusor
- BOTOX 50 U: botulinum toxin Type A 50 U injection on Day 1 into detrusor
- BOTOX 100 U: botulinum toxin Type A 100 U injection on Day 1 into detrusor
- BOTOX 150 U: botulinum toxin Type A 150 U injection on Day 1 into detrusor
- BOTOX 200 U: botulinum toxin Type A 200 U injection on Day 1 into detrusor
- BOTOX 300 U: botulinum toxin Type A 300 U injection on Day 1 into detrusor
Period: Overall Study
Arm/Group | Placebo | BOTOX 50 U | BOTOX 100 U | BOTOX 150 U | BOTOX 200 U | BOTOX 300 U
Started | 44 | 57 | 54 | 49 | 53 | 56
Completed | 37 | 50 | 48 | 40 | 47 | 50
Not Completed | 7 | 7 | 6 | 9 | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BOTOX 50 U | BOTOX 100 U | BOTOX 150 U | BOTOX 200 U | BOTOX 300 U | Total
Number analyzed (Participants) | 44 | 57 | 54 | 49 | 53 | 56 | 313
Age, Customized [Number; unit: participants]
  <45 years | 7 | 9 | 6 | 8 | 6 | 6 | 42
  45-64 years | 24 | 27 | 25 | 27 | 21 | 29 | 153
  65-74 years | 6 | 13 | 16 | 12 | 20 | 15 | 82
  >=75 years | 7 | 8 | 7 | 2 | 6 | 6 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 53 | 50 | 47 | 46 | 52 | 288
  Male | 4 | 4 | 4 | 2 | 7 | 4 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Urinary Urge Incontinence Episodes
Description: Mean number of urinary urge incontinence episodes measured over a 7-day diary prior to week 12. Urinary urge incontinence is defined as urinary leakage associated with a strong desire to urinate.
Time Frame: Baseline, Week 2, Week 6, Week 12
Population: Intent to Treat
Measure: Number; unit: episodes
Arm/Group | Placebo | BOTOX 50 U | BOTOX 100 U | BOTOX 150 U | BOTOX 200 U | BOTOX 300 U
Number analyzed (Participants) | 44 | 57 | 54 | 49 | 53 | 56
episodes
  Baseline | 32.5 | 30.3 | 27.8 | 28.3 | 24.1 | 26.8
  Week 2 | -17.3 | -20.0 | -18.6 | -20.8 | -16.8 | -18.6
  Week 6 | -18.2 | -21.2 | -19.9 | -23.4 | -20.0 | -18.8
  Week 12 | -17.4 | -20.7 | -18.4 | -23.0 | -19.6 | -19.4

2. Secondary Outcome: Change in Number of Micturitions
Description: Mean number of micturitions measured over a 7 day diary prior to each visit. Micturation is defined as urinating into the toilet.
Time Frame: Baseline, Week 2, Week 6, Week 12
Population: Intent to Treat
Measure: Number; unit: micturitions
Arm/Group | Placebo | BOTOX 50 U | BOTOX 100 U | BOTOX 150 U | BOTOX 200 U | BOTOX 300 U
Number analyzed (Participants) | 44 | 57 | 54 | 49 | 53 | 56
micturitions
  Baseline | 73.3 | 76.3 | 80.3 | 76.5 | 76.7 | 75.6
  Week 2 | -6.5 | -10.0 | -12.5 | -9.8 | -7.2 | -9.2
  Week 6 | -9.4 | -15.2 | -22.9 | -17.0 | -18.9 | -19.9
  Week 12 | -8.3 | -15.3 | -21.7 | -18.8 | -19.7 | -21.2

3. Secondary Outcome: Change in Number of Nocturia Episodes
Description: Mean number of nocturia episodes measured over a 7 day diary prior to each visit. A nocturia episode is a void (urinating into the toilet) that interrupts one's sleep.
Time Frame: Baseline, Week 12
Population: Intent to Treat
Measure: Number; unit: episodes
Arm/Group | Placebo | BOTOX 50 U | BOTOX 100 U | BOTOX 150 U | BOTOX 200 U | BOTOX 300 U
Number analyzed (Participants) | 44 | 57 | 54 | 49 | 53 | 56
episodes
  Baseline | 12.3 | 12.2 | 13.9 | 17.9 | 12.2 | 14.9
  Week 12 | -0.3 | -2.5 | -4.1 | -6.5 | -3.8 | -7.0

4. Secondary Outcome: Maximum Cystometric Capacity (MCC) by Urodynamic Measurements
Description: Maximum Cystometric Capacity (maximum volume that the bladder can hold) measured in mean milliliters
Time Frame: Baseline, Week 12
Population: Intent to Treat
Measure: Number; unit: milliliters
Arm/Group | Placebo | BOTOX 50 U | BOTOX 100 U | BOTOX 150 U | BOTOX 200 U | BOTOX 300 U
Number analyzed (Participants) | 44 | 57 | 54 | 49 | 53 | 56
milliliters
  Baseline | 267.1 | 262.9 | 255.0 | 258.4 | 280.1 | 271.7
  Week 12 | 49.5 | 50.0 | 71.0 | 101.7 | 91.5 | 130.8

5. Secondary Outcome: Incontinence Quality of Life Instrument (I-QOL)
Description: Measured on 3 domains; a 5-point scale (1-5) for each domain. Sum of the domain scores is normalized to a scale of 0-100 (100 = no impact of incontinence on daily activities, 0 = maximum impact of incontinence on daily activities). Mean scores presented.
Time Frame: Baseline, Week 2, Week 6, Week 12
Population: Intent to Treat
Measure: Number; unit: Units on a scale
Arm/Group | Placebo | BOTOX 50 U | BOTOX 100 U | BOTOX 150 U | BOTOX 200 U | BOTOX 300 U
Number analyzed (Participants) | 44 | 57 | 54 | 49 | 53 | 56
Units on a scale
  Baseline | 35.9 | 32.3 | 34.3 | 30.5 | 32.0 | 34.5
  Week 2 | 14.8 | 21.1 | 28.1 | 29.5 | 26.7 | 31.6
  Week 6 | 16.3 | 30.6 | 32.1 | 37.2 | 34.5 | 41.6
  Week 12 | 17.9 | 29.8 | 32.9 | 35.2 | 37.1 | 39.7

6. Post Hoc Outcome: Percentage of Patients With 100% Reduction From Baseline of Urinary Urge Incontinence Episodes
Description: Measured by the 7 day diary preceding each visit. Urinary urge incontinence is defined as urinary leakage associated with a strong desire to urinate.
Time Frame: Baseline, Week 2, Week 6, Week 12, Week 18, Week 24, Week 30, Week 36
Population: Intent to Treat
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | BOTOX 50 U | BOTOX 100 U | BOTOX 150 U | BOTOX 200 U | BOTOX 300 U
Number analyzed (Participants) | 44 | 57 | 54 | 49 | 53 | 56
Percentage of patients
  Week 2 | 11.4 | 12.3 | 27.8 | 26.5 | 28.3 | 44.6
  Week 6 | 18.2 | 24.6 | 44.4 | 49.0 | 49.1 | 55.4
  Week 12 | 15.9 | 29.8 | 37.0 | 40.8 | 50.9 | 57.1
  Week 18 | 13.6 | 26.3 | 38.9 | 44.9 | 39.6 | 46.4
  Week 24 | 13.6 | 28.1 | 27.8 | 42.9 | 54.7 | 53.6
  Week 30 | 18.2 | 21.1 | 35.2 | 28.6 | 41.5 | 46.4
  Week 36 | 11.4 | 15.8 | 33.3 | 36.7 | 32.1 | 42.9

ADVERSE EVENTS:
Description: The Safety Population is defined as all randomized patients who received treatment and was used to analyze Serious Adverse Events and Adverse Events.
Arm/Group | Placebo | BOTOX 50 U | BOTOX 100 U | BOTOX 150 U | BOTOX 200 U | BOTOX 300 U
Serious Adverse Events (participants affected / at risk) | 5 | 9 | 5 | 7 | 4 | 4
Other Adverse Events (participants affected / at risk) | 33 | 44 | 44 | 39 | 44 | 46
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Placebo | BOTOX 50 U | BOTOX 100 U | BOTOX 150 U | BOTOX 200 U | BOTOX 300 U
Atrial Fibrillation (Cardiac disorders) | 0/43 | 1/56 | 0/55 | 0/50 | 1/52 | 0/55
Angina pectoris (Cardiac disorders) | 0/43 | 0/56 | 0/55 | 1/50 | 0/52 | 0/55
Coronary artery disease (Cardiac disorders) | 0/43 | 0/56 | 0/55 | 1/50 | 0/52 | 0/55
Cardiac failure congestive (Cardiac disorders) | 0/43 | 0/56 | 1/55 | 0/50 | 0/52 | 0/55
Ileus (Gastrointestinal disorders) | 0/43 | 0/56 | 0/55 | 0/50 | 0/52 | 1/55
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0/43 | 0/56 | 0/55 | 0/50 | 1/52 | 0/55
Impaired gastric emptying (Gastrointestinal disorders) | 0/43 | 1/56 | 0/55 | 0/50 | 0/52 | 0/55
Cholelithiasis (Hepatobiliary disorders) | 0/43 | 0/56 | 0/55 | 0/50 | 1/52 | 0/55
Diverticulitis (Infections and infestations) | 0/43 | 1/56 | 0/55 | 0/50 | 0/52 | 1/55
Bacterial pyelonephritis (Infections and infestations) | 0/43 | 1/56 | 0/55 | 0/50 | 0/52 | 0/55
Urinary tract infection (Infections and infestations) | 0/43 | 1/56 | 0/55 | 0/50 | 0/52 | 0/55
Herpes ophthalmic (Infections and infestations) | 1/43 | 0/56 | 0/55 | 0/50 | 0/52 | 0/55
Skeletal injury (Injury, poisoning and procedural complications) | 0/43 | 0/56 | 0/55 | 0/50 | 1/52 | 0/55
Concussion (Injury, poisoning and procedural complications) | 1/43 | 0/56 | 0/55 | 0/50 | 0/52 | 0/55
Hip Fracture (Injury, poisoning and procedural complications) | 1/43 | 0/56 | 0/55 | 0/50 | 0/52 | 0/55
Dehydration (Metabolism and nutrition disorders) | 0/43 | 1/56 | 0/55 | 0/50 | 0/52 | 1/55
Diabetes mellitus (Metabolism and nutrition disorders) | 0/43 | 0/56 | 0/55 | 1/50 | 0/52 | 0/55
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/43 | 0/56 | 2/55 | 1/50 | 0/52 | 0/55
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0/43 | 0/56 | 1/55 | 0/50 | 0/52 | 0/55
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1/43 | 0/56 | 0/55 | 0/50 | 0/52 | 0/55
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/43 | 0/56 | 0/55 | 2/50 | 0/52 | 2/55
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/43 | 0/56 | 0/55 | 1/50 | 0/52 | 0/55
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/43 | 0/56 | 1/55 | 0/50 | 0/52 | 0/55
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/43 | 1/56 | 0/55 | 0/50 | 0/52 | 0/55
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/43 | 0/56 | 0/55 | 0/50 | 0/52 | 0/55
Squamos cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/43 | 0/56 | 0/55 | 0/50 | 0/52 | 0/55
Convulsion (Nervous system disorders) | 0/43 | 0/56 | 0/55 | 0/50 | 0/52 | 1/55
Headache (Nervous system disorders) | 0/43 | 0/56 | 0/55 | 1/50 | 0/52 | 0/55
Syncope (Nervous system disorders) | 0/43 | 0/56 | 0/55 | 1/50 | 0/52 | 0/55
Ischaemic stroke (Nervous system disorders) | 0/43 | 1/56 | 0/55 | 0/50 | 0/52 | 0/55
Normal pressure hydrocephalus (Nervous system disorders) | 1/43 | 0/56 | 0/55 | 0/50 | 0/52 | 0/55
Schizophrenia, undifferentiated type (Psychiatric disorders) | 0/43 | 0/56 | 0/55 | 0/50 | 1/52 | 0/55
Cystitis noninfective (Renal and urinary disorders) | 0/43 | 0/56 | 1/55 | 0/50 | 0/52 | 0/55
Urinary retention (Renal and urinary disorders) | 0/43 | 0/56 | 1/55 | 0/50 | 0/52 | 0/55
Ovarian cyst (Reproductive system and breast disorders) | 0/43 | 1/56 | 0/55 | 0/50 | 0/52 | 0/55
Hypertension (Vascular disorders) | 0/43 | 0/56 | 0/55 | 0/50 | 1/52 | 0/55
Hypotension (Vascular disorders) | 0/43 | 0/56 | 0/55 | 1/50 | 0/52 | 0/55
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Placebo | BOTOX 50 U | BOTOX 100 U | BOTOX 150 U | BOTOX 200 U | BOTOX 300 U
Urinary tract infection (Infections and infestations) | 7/43 | 19/56 | 20/55 | 22/50 | 25/52 | 19/55
Upper respiratory tract infection (Infections and infestations) | 2/43 | 3/56 | 3/55 | 4/50 | 2/52 | 5/55
Bronchitis (Infections and infestations) | 0/43 | 2/56 | 3/55 | 0/50 | 2/52 | 3/55
Nasopharyngitis (Infections and infestations) | 1/43 | 1/56 | 6/55 | 1/50 | 2/52 | 2/55
Influenza (Infections and infestations) | 0/43 | 1/56 | 3/55 | 3/50 | 5/52 | 1/55
Lower respiratory tract infection (Infections and infestations) | 0/43 | 1/56 | 3/55 | 2/50 | 0/52 | 1/55
Sinusitis (Infections and infestations) | 2/43 | 5/56 | 2/55 | 1/50 | 0/52 | 1/55
Urinary retention (Renal and urinary disorders) | 1/43 | 5/56 | 10/55 | 14/50 | 12/52 | 14/55
Bladder pain (Renal and urinary disorders) | 1/43 | 1/56 | 0/55 | 4/50 | 1/52 | 2/55
Pollakiuria (Renal and urinary disorders) | 0/43 | 4/56 | 1/55 | 1/50 | 0/52 | 2/55
Dysuria (Renal and urinary disorders) | 5/43 | 7/56 | 1/55 | 4/50 | 6/52 | 1/55
Renal cyst (Renal and urinary disorders) | 2/43 | 2/56 | 0/55 | 1/50 | 3/52 | 1/55
Haematuria (Renal and urinary disorders) | 6/43 | 5/56 | 0/55 | 2/50 | 1/52 | 0/55
Diarrhoea (Gastrointestinal disorders) | 1/43 | 5/56 | 2/55 | 1/50 | 3/52 | 2/55
Nausea (Gastrointestinal disorders) | 4/43 | 1/56 | 4/55 | 0/50 | 2/52 | 1/55
Abdominal pain (Gastrointestinal disorders) | 4/43 | 3/56 | 1/55 | 0/50 | 0/52 | 1/55
White blood cells urine positive (Investigations) | 2/43 | 1/56 | 4/55 | 1/50 | 3/52 | 2/55
Residual urine volume (Investigations) | 0/43 | 3/56 | 1/55 | 3/50 | 4/52 | 1/55
Blood urine present (Investigations) | 3/43 | 1/56 | 1/55 | 0/50 | 0/52 | 1/55
Back pain (Musculoskeletal and connective tissue disorders) | 5/43 | 1/56 | 3/55 | 1/50 | 0/52 | 3/55
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2/43 | 0/56 | 3/55 | 1/50 | 0/52 | 3/55
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/43 | 0/56 | 2/55 | 2/50 | 4/52 | 1/55
Dizziness (Nervous system disorders) | 1/43 | 3/56 | 5/55 | 0/50 | 0/52 | 3/55
Headache (Nervous system disorders) | 2/43 | 1/56 | 0/55 | 2/50 | 3/52 | 1/55
Sciatica (Nervous system disorders) | 3/43 | 0/56 | 1/55 | 1/50 | 0/52 | 0/55
Rash (Skin and subcutaneous tissue disorders) | 1/43 | 2/56 | 0/55 | 1/50 | 0/52 | 3/55
Ovarian cyst (Reproductive system and breast disorders) | 0/43 | 3/56 | 2/55 | 0/50 | 0/52 | 0/55
Cough (Respiratory, thoracic and mediastinal disorders) | 0/43 | 0/56 | 3/55 | 1/50 | 1/52 | 1/55
Hypertension (Vascular disorders) | 2/43 | 1/56 | 1/55 | 2/50 | 3/52 | 1/55
Depression (Psychiatric disorders) | 1/43 | 1/56 | 3/55 | 1/50 | 1/52 | 1/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less